CLINICAL TRIAL: NCT02948881
Title: A One Year, Parallel, Placebo-controlled, Double-blind, Randomized Study to Assess the Effect of Monthly 150mg Oral Ibandronate Dosing Versus Placebo on Bone Quality and Strength at the Proximal Femur in Women With Osteoporosis
Brief Title: A Study To Assess The Quality Of Bone In Patients Taking Oral Ibandronate Versus Placebo
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BON103593
Record Dates: First submitted 2016-10-27; First posted 2016-10-31 (Estimated); Last update posted 2016-10-31 (Estimated); Status verified 2016-10

CONDITIONS: Osteoporosis
Keywords: Osteoporosis; bisphosphonates; bone
MeSH Terms: conditions — Osteoporosis | interventions — Ibandronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: ibandronate

SUMMARY:
The purpose of this study is to estimate the effect of oral Boniva (ibandronate sodium)taken once monthly versus placebo on bone quality and strength at the hip at one year.

ELIGIBILITY:
Inclusion criteria:

* Ambulatory, postmenopausal women who are diagnosed with osteoporosis.
* Must be able to stand or sit upright for at least 60 minutes and swallow a tablet whole.

Exclusion criteria:

* Have been treated with other bisphosphonates or using chronic steroids within the past 6 months.
* Have a history of major upper GI diseases or have severe kidney dysfunction.
* Have a spine fracture (identified on x-ray).

Ages: 55 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2005-08; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Bone quality and strength at the hip by characterizing changes in trabecular and cortical bone quality using Volumetric Quantitative Computed Tomography (vQCT) and novel imaging analysis methods, including a subset of bone biopsies for one year. | 1 Year

SECONDARY OUTCOMES:
Relationship between biomarkers and changes in bone quality for one year. | 1 Year

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (14):
- United States (14):
  - GSK Investigational Site, Upland, California
  - GSK Investigational Site, Boulder, Colorado
  - GSK Investigational Site, Lakewood, Colorado
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, West Palm Beach, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Decatur, Georgia
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, Bangor, Maine
  - GSK Investigational Site, Bathesda, Maryland
  - GSK Investigational Site, Flint, Michigan
  - GSK Investigational Site, Albuquerque, New Mexico
  - GSK Investigational Site, West Haverstraw, New York
  - GSK Investigational Site, Duncansville, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: BON103593 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: BON103593 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: BON103593 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: BON103593 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: BON103593 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: BON103593 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: BON103593 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register